CLINICAL TRIAL: NCT03069196
Title: A Study to Assess Prevalence and Incidence of Long-term Complications of Type 1 Diabetes in a Tertiary Clinic in Pune.
Brief Title: Prevalence and Incidence of Complications of Type One Diabetes in PUne At a Tertiary Care CentRE
Acronym: PICTURE
Status: Active, not recruiting | Type: Observational
Sponsor: Kem Hospital, Pune, India (Other)
Responsible Party: Principal Investigator, Dr. Chittaranjan S Yajnik, Professor Dr., King Edward Memorial Hospital
Other Study IDs: PhD 19
Record Dates: First submitted 2017-02-16; First posted 2017-03-03 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Prevalence; Incidence; Type 1 diabetes and its Micro-vascular complications; Type 1 diabetes and its Macro-vascular complications; Type 1 Diabetes and its complications in India
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For future biochemical tests : Plasma, Serum and Urine samples are stored. To do DNA extraction at a later stage Packed cells are stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Due to early diagnosis (<20yrs of age) of Type 1 Diabetes, patients face longer duration of disease and greater glycemic exposure which makes them more vulnerable towards chronic complications. The aim of this study is to investigate the prevalence and incidence of micro and macro-vascular, pulmonary complications and patterns of growth failure in approximately 500 Type 1 Diabetes patients enrolled at Diabetes Unit, King Edward Memorial Hospital Research Centre. Then follow up of 100 participants who are above 15 years of age at baseline will be done after 2 years to document incidence and progression of complications. This will contribute in assessing the public health burden of complications of Type 1 Diabetes.

Factors associated with prevalence of complications will be investigated. This risk factor analysis could aid in further modifying current prevention and treatment recommendations of these complications. Results of this study could modify current clinical practice.

DETAILED DESCRIPTION:
BACKGROUND & RATIONALE OF THE STUDY:

Type 1 Diabetes (T1D) is characterized by progressive destruction of insulin secreting pancreatic β-cells. The commonest mechanism involves autoimmunity to components of β-cells. As per International Diabetes Federation report 2013, India houses 67,700 children (<15yrs) with T1D. It also states an approximate figure of 10,900 newly diagnosed T1D children (<15yrs) per year. India accounts for highest number of children with T1D in South East Asian Region. Karnataka Diabetes Registry of T1D patients (1995 to 2008) reported an incidence of 3.8per 100,000 persons in India which is less when compared to Europe and other Western countries. Same study also reported that there is a huge gap between international standard of care and practice in India and that majority of T1D patients don't attain their glycemic targets.

Despite such unfavorable statistics, T1D does not receive adequate attention in terms of clinical and epidemiological research, achieving standards of practice and training of Medical practitioners. Many a times, it is also quoted as "Poor Cousin of Type 2 Diabetes".

A salient feature of T1D is its early onset and diagnosis (<20yrs of age) compared to type 2 diabetes. Consequently patients face longer duration of disease and greater glycemic exposure by the time they reach productive age and suffer chronic complications which are broadly classified into:

1. Microvascular (retinopathy, neuropathy, and nephropathy) and
2. Macrovascular [coronary artery disease (CAD), cerebrovascular disease (CVD), peripheral vascular disease (PVD)] .

These complications contribute to poor quality, substantial morbidity and premature mortality during prime years of life and premature death in T1D patients.

Limited studies are available from India on micro and macro-vascular complication of T1D.

Previous studies have detected that atherosclerotic process is accelerated in T1D population and western studies demonstrated a premature thickening of arterial Intima Media Thickness (IMT) within a short disease duration. Schuyler et al in 1976 for the first time suggested pulmonary complications among T1D. Since then limited attention has been given to lung as a target organ of diabetes even when lungs have a large vascular network. Studies have reported peripheral airway dysfunction and restrictive impairment of lung function even in the absence of smoking, allergies and other causes of airflow destruction among T1D patients. Screening for pulmonary complications among patients with T1D is currently not included in routine clinical settings. Growth parameters like standing height, weight are important indicators of a child's overall health and T1D patients are at an increased risk of developing growth failure. This is due to the role of insulin as a main regulator of Growth Hormone/Insulin Growth Factors (GH/IGF) axis and presence of portal insulin insufficiency among T1D patients. A recent study from Pune reported compromised growth in diabetic children when compared to matched controls. Impaired pre-pubertal and pubertal growth in children and adolescents has been reported in many studies. Factors like gender, age at diagnosis, puberty, metabolic control, insulin regime all affect growth. Bonfig et al 2012 observed a negative association between degree of metabolic control and impaired growth.

Risk factors for complications of T1D have been studied in Western population. Most of them report duration of disease, hyperglycemia, hypertension and dyslipidemia as predictors for micro and macro-vascular complications. But surprisingly "the 50-yr Medalist study" found no association of glycemic control with prevalence of micro-vascular complications.

Research Gap:

The public health burden of T1D is increasing in India and cannot be ignored. Studies assessing long-term complications of T1D from India are limited. They have relatively small sample size, are cross-sectional and retrospective in design. Incidence and progression of these complications has not been reported from India.Prevalence and progression of pulmonary complication among T1D patients has not been studied. Growth data in T1D patients is also limited and will benefit from our study.

Aims and Objectives :

Aim: This thesis will investigate prevalence; incidence and progression of micro-vascular, macro-vascular, pulmonary complications and growth failure among T1D patients in a clinic setting (specialty Diabetes Unit).

1. OBJECTIVE 1 : To determine the prevalence of long-term complications among T1D patients.
2. OBJECTIVE 2 : To determine the impact of factors like age, socio-economic status, body mass index (BMI), body fat (adiposity), duration of disease and glycemic control on the prevalence of complications.
3. OBJECTIVE 3 :To document clinical progression of these complications in duration of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes with a duration of diabetes more than 1 year.
* Willingness to participate in the study and sign the consent form.
* Age : all age groups
* Gender : Both

Exclusion Criteria:

* Other forms of diabetes like Type 2 Diabetes, Gestational Diabetes, Fibro Calculus Pancreatic Disease (FCPD), Mature Onset of Diabetes in Young (MODY) etc.
* People with acute stages of diseases like pneumonia after being treated for the condition.
* Advanced end stage conditions like Cancer etc.
* Pregnant and lactating women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes those people who have been clinically diagnosed with Type 1 Diabetes. These participants will be selected from those enrolled at Diabetes Unit, KEMHRC, Pune, India.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Micro-vascular Complications. | Assessed in one day, approximately.
  Following tests will be performed for micro-vascular complications :
  1. RETINOPATHY: Retina scan images
  2. NEPHROPATHY:Urine Albumin : Creatinine ratio), Serum Creatinine, estimated glomerular filtration rate (eGFR)
  3. NEUROPATHY : Michigan Neuropathy Screening Instrument (MNSI) and Biothesiometer.
  4. Pulmonary : Spirometry
  Prevalence will be reported as percentage i.e. number of cases divided by total number of study participants , multiplied by 100.
Prevalence of Macro-vascular Complications. | Assessed in one day, approximately.
  Following tests will be performed for macro-vascular complications :
  1. Cardio-Vascular Disease :Blood pressure, Biochemical tests: Lipid Profile [Triglycerides, Cholesterol (HDL, LDL, total)] and ECG (Electrocardiogram > 15 years of age)
  2. Peripheral Vascular Disease : Ankle Brachial Index by Periscope
  Prevalence will be reported as percentage i.e. number of cases divided by total number of study participants , multiplied by 100.
Prevalence of Growth Complications. | Assessed in one day, approximately.
  Whole body Anthropometry and Pubertal staging by Tanner's method.
Incidence of Micro-vascular, Macro-Vascular and Pulmonary Complications. | Assessed in one day, approximately.
  Same tools as listed for primary objective 1 will be utilised for measuring incidence of these complications.
  - Incidence will be reported as number of new cases per year.
Progression of Micro-vascular, Macro-Vascular and Pulmonary Complications. | Assessed in one day, approximately.
  Same tools as listed for primary objective 1 will be utilised for measuring incidence of these complications.
  - Incidence will be reported as number of new cases per year.

SECONDARY OUTCOMES:
Association of Risk factors with prevalence of complications. | All this data will be collected at the time of primary objective 1 i.e. in one day.
  Risk factors are : BMI, Body fat, duration of disease, glycemic control (HbA1C), clinical history, family history, socio-economic status, Lifestyle related: Diet, Physical Activity and substance abuse, Body Composition : whole body Anthropometry and Dual Energy X-ray absorptiometry (DXA).
  Risk factors will be used for multivariate analysis with the incidence and prevalence rates, also to report relative risks.

CONTACTS AND LOCATIONS:
Overall Officials: Chittaranjan Yajnik, MD, FRCP, Principal Investigator — KEMHRC
Locations (1):
- Diabetes Unit, Kem Hospital Research Centre, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andersson K, Fuxe K, Eneroth P, Mascagni F, Agnati LF. Effects of acute intermittent exposure to cigarette smoke on catecholamine levels and turnover in various types of hypothalamic DA and NA nerve terminal systems as well as on the secretion of adenohypophyseal hormones and corticosterone. Acta Physiol Scand. 1985 Jun;124(2):277-85. doi: 10.1111/j.1748-1716.1985.tb07662.x. PMID 2861716
- [Background] Groenendijk-Huijbers MM, Burggraaff JM. Experimental studies on the capability of embryonic and young chick testes to regress embryonic chick oviducts. Anat Anz. 1974;135(1-2):43-6. No abstract available. PMID 4413385
- [Background] Hugues CJ, Asmar RG, London GM, Safar ME. Age- and sex-related changes in the ratio between ankle and brachial systolic pressure in normal subjects. Angiology. 1988 Mar;39(3 Pt 1):219-26. doi: 10.1177/000331978803900303. PMID 3354924
- [Background] Walsh MG, Zgibor J, Borch-Johnsen K, Orchard TJ; DiaMond Investigators. A multinational comparison of complications assessment in type 1 diabetes: the DiaMond substudy of complications (DiaComp) level 2. Diabetes Care. 2004 Jul;27(7):1610-7. doi: 10.2337/diacare.27.7.1610. PMID 15220236
- [Background] Pickup, John C and Williams, Gareth, MD Textbook of diabetes (3rd ed). Blackwell Science, Malden, Mass. ; Oxford, U.K, 2003.
- [Background] Patterson C, Guariguata L, Dahlquist G, Soltesz G, Ogle G, Silink M. Diabetes in the young - a global view and worldwide estimates of numbers of children with type 1 diabetes. Diabetes Res Clin Pract. 2014 Feb;103(2):161-75. doi: 10.1016/j.diabres.2013.11.005. Epub 2013 Dec 1. PMID 24331235
- [Background] Amutha A, Thai K, Vishwanathan M. Childhood and Adolescent ONset Type 1 Diabetes in India. MGM Journal of Medical Sciences. 2013; 1(1): p. 46-53.
- [Background] Unnikrishnan AG, Bhatia E, Bhatia V, Bhadada SK, Sahay RK, Kannan A, Kumaravel V, Sarma D, Ganapathy B, Thomas N, John M, Jayakumar RV, Kumar H, Nair V, Sanjeevi CB. Type 1 diabetes versus type 2 diabetes with onset in persons younger than 20 years of age. Ann N Y Acad Sci. 2008 Dec;1150:239-44. doi: 10.1196/annals.1447.056. PMID 19120303
- [Background] Billow A, Anjana RM, Ngai M, Amutha A, Pradeepa R, Jebarani S, Unnikrishnan R, Michael E, Mohan V. Prevalence and clinical profile of metabolic syndrome among type 1 diabetes mellitus patients in southern India. J Diabetes Complications. 2015 Jul;29(5):659-64. doi: 10.1016/j.jdiacomp.2015.03.014. Epub 2015 Apr 6. PMID 25899474
- [Background] Ramachandran A, Snehalatha C, Sasikala R, Satyavani K, Vijay V. Vascular complications in young Asian Indian patients with type 1 diabetes mellitus. Diabetes Res Clin Pract. 2000 Apr;48(1):51-6. doi: 10.1016/s0168-8227(99)00134-5. PMID 10704700
- [Background] Laing SP, Swerdlow AJ, Slater SD, Burden AC, Morris A, Waugh NR, Gatling W, Bingley PJ, Patterson CC. Mortality from heart disease in a cohort of 23,000 patients with insulin-treated diabetes. Diabetologia. 2003 Jun;46(6):760-5. doi: 10.1007/s00125-003-1116-6. Epub 2003 May 28. PMID 12774166
- [Background] Dawson SI, Willis J, Florkowski CM, Scott RS. Cause-specific mortality in insulin-treated diabetic patients: a 20-year follow-up. Diabetes Res Clin Pract. 2008 Apr;80(1):16-23. doi: 10.1016/j.diabres.2007.10.034. Epub 2008 Mar 7. PMID 18329124
- [Background] Singh TP, Groehn H, Kazmers A. Vascular function and carotid intimal-medial thickness in children with insulin-dependent diabetes mellitus. J Am Coll Cardiol. 2003 Feb 19;41(4):661-5. doi: 10.1016/s0735-1097(02)02894-2. PMID 12598080
- [Background] Stakos DA, Schuster DP, Sparks EA, Wooley CF, Osei K, Boudoulas H. Cardiovascular effects of type 1 diabetes mellitus in children. Angiology. 2005 May-Jun;56(3):311-7. doi: 10.1177/000331970505600311. PMID 15889199
- [Background] Schuyler MR, Niewoehner DE, Inkley SR, Kohn R. Abnormal lung elasticity in juvenile diabetes mellitus. Am Rev Respir Dis. 1976 Jan;113(1):37-41. doi: 10.1164/arrd.1976.113.1.37. PMID 1247213
- [Background] Pitocco D, Fuso L, Conte EG, Zaccardi F, Condoluci C, Scavone G, Incalzi RA, Ghirlanda G. The diabetic lung--a new target organ? Rev Diabet Stud. 2012 Spring;9(1):23-35. doi: 10.1900/RDS.2012.9.23. Epub 2012 May 10. PMID 22972442
- [Background] Goldman MD. Lung dysfunction in diabetes. Diabetes Care. 2003 Jun;26(6):1915-8. doi: 10.2337/diacare.26.6.1915. No abstract available. PMID 12766133
- [Background] van den Borst B, Gosker HR, Zeegers MP, Schols AM. Pulmonary function in diabetes: a metaanalysis. Chest. 2010 Aug;138(2):393-406. doi: 10.1378/chest.09-2622. Epub 2010 Mar 26. PMID 20348195
- [Background] Giannini C, Mohn A, Chiarelli F. Growth abnormalities in children with type 1 diabetes, juvenile chronic arthritis, and asthma. Int J Endocrinol. 2014;2014:265954. doi: 10.1155/2014/265954. Epub 2014 Feb 4. PMID 24648838
- [Background] Khadilkar VV, Parthasarathy LS, Mallade BB, Khadilkar AV, Chiplonkar SA, Borade AB. Growth status of children and adolescents with type 1 diabetes mellitus. Indian J Endocrinol Metab. 2013 Nov;17(6):1057-60. doi: 10.4103/2230-8210.122623. PMID 24381884
- [Background] Bonfig W, Kapellen T, Dost A, Fritsch M, Rohrer T, Wolf J, Holl RW; Diabetes Patienten Verlaufsdokumentationssystem Initiative of the German Working Group for Pediatric Diabetology and the German Bundesministerium fur Bildung und Forschung Competence Net for Diabetes Mellitus. Growth in children and adolescents with type 1 diabetes. J Pediatr. 2012 Jun;160(6):900-3.e2. doi: 10.1016/j.jpeds.2011.12.007. Epub 2012 Jan 11. PMID 22244464
- [Background] Grauslund J, Jorgensen TM, Nybo M, Green A, Rasmussen LM, Sjolie AK. Risk factors for mortality and ischemic heart disease in patients with long-term type 1 diabetes. J Diabetes Complications. 2010 Jul-Aug;24(4):223-8. doi: 10.1016/j.jdiacomp.2009.05.003. Epub 2009 Jul 3. PMID 19577486
- [Background] Keenan HA, Costacou T, Sun JK, Doria A, Cavellerano J, Coney J, Orchard TJ, Aiello LP, King GL. Clinical factors associated with resistance to microvascular complications in diabetic patients of extreme disease duration: the 50-year medalist study. Diabetes Care. 2007 Aug;30(8):1995-7. doi: 10.2337/dc06-2222. Epub 2007 May 16. No abstract available. PMID 17507696